CLINICAL TRIAL: NCT04955106
Title: Evaluation of the Relability and Validity of Device for the Screening of Early Pressure Ulcer in Hospitalization High-risk Patient, the Sub Epidermal Moisture During a Monocebtric Study
Brief Title: Evaluation of the Sub Epidermal Moisture a Device for the Screening of Pressure Ulcer (RELIASEM)
Acronym: RELIASEM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arjo France (Industry)
Collaborators: Pôle Saint Hélier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021-A00458-33
Record Dates: First submitted 2021-06-24; First posted 2021-07-08 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Preventive Care

STUDY DESIGN:
Intervention Model Description: The SEM Scanner is placed on three skin areas (left heel, right heel and sacrum). It measures the moisture of the subcutaneous tissues. If returns a figure wich induces a classification
  * negative = value <0.6 no risk, the figure is displayed in green
  * positive = value ≥0.6 proven risk, the figure is displayed in orange
  For each patient 3 measurements will be performed. Two of them will have been trained in the use of the SEM Scanner, whereas the others will be novice
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sample for reliability (Other): Reliability and validity of SEM Scanner : intra rater, inter rater and inter novice/trained 8(2 trained rater, 2 novice rater, each one performed twice)measured will be performed on each patient.
  Interventions: Diagnostic Test: SEM Scanner

INTERVENTIONS:
Diagnostic Test: SEM Scanner — They will perform 2 sets of 3 measures (1 on sacrum, 1 on the right heel and 1 on the left heel)for each patients

SUMMARY:
The device that is the subject of this investigation is a diagnostic tool to detect the among of fluid in hypodermis to help to prevent the formation of pressure injuries. The Sub Epidermal Moister(SEM) Scanner, is a non invasive portable medical device use to complet the clinical jugement of clinician

DETAILED DESCRIPTION:
The device that is the subject of this investigation is a diagnostic tool to detect the among of fluid in hypodermis to help to prevent the formation of pressure injuries. The Sub Epidermal Moister(SEM) Scanner, is a non invasive portable medical device use to complet the clinical jugement of clinician.

The study "RELIASEM" will study hospitalized patients with high risk of Pressure Injurieswith the next conditions:

For each patient 14 mesures: 6 on the sacrum, 4 on the right heel and 4 on the left heel. This set of measure will be realized 2 timesby 4 different evaluator. To will have been trained in the use of the SEM Scanner where as the other will be novice.

The main objective of this study is to determine on a risk population the intra- and inter-examiner reliability of the SEM Scanner

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18
* Taken the full-hospital care in physical and rehabilitation Medicine
* Patient affiliated with a social security scheme
* In the case of curatorship, patient have read the patient information document and given his consent free and informed, in the presence of his/her curator
* In the case of guardianship, legal representative have to had read the legal representative information document for major placed under legal protection (under guardianship) and given his consent free and informed for the person for whom he is responsible (if the patient is agree),

Exclusion Criteria:

* Patient who objected his opposition during the exam
* Patient who have one or more presure ulcer on at list one of the measuring area
* Patient who has had a lower limb amputation
* Pregnant, post natal period or breastfeeding women,
* Person deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the reliability of the SEM Scanner on a population in a rehabilitation center (experienced vs experienced) | immediately after the intervention
  We will calculate the intra-class correlation coefficient (ICC) intra- and inter-evaluator (experienced vs experienced)
Evaluation of the validity of the SEM Scanner on at risk population | immediately after the intervention
  Intra-class correlation coefficient is the correlation coefficient between SEM Scanner measure and the norton scare
Evaluation of the validity of the SEM Scanner on at risk population | During the evaluation 1 day assessed
  The Norton scale will be used by the study :Norton ≥ 18 low or without risk, 14< Norton <18 medium risk, 12≤ Norton ≤14 high risk, Norton < 12 very high risk

SECONDARY OUTCOMES:
valuation of the reliability of the SEM Scanner on a population at risk (experienced vs novice/ novice vs novice) will be calculated | immediately after the intervention
  The intra-class correlation coefficient (ICC) intra- and inter- evaluator (experienced vs novice/novice vs novice) will be calculated
Receiver Operating Characteristics (ROC)curve: Area under the Curve (AUC) | immediately after the intervention
  AUC of the SEM Scanner for every cut of scores of the Norton score

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Gallien, Doctor, Principal Investigator — Pôle Saint Hélier
Locations (1):
- Pole Saint-Hélier, Rennes, Brittany Region, France